CLINICAL TRIAL: NCT06273085
Title: Intensive Education Versus Usual Education of Patients for Improving Guideline Directed Medical Therapy (GDMT) Prescription in Heart Failure With Reduced Ejection Fraction- A Randomized Controlled Trial
Brief Title: Intensive Education Versus Usual Education of Patients for Improving Guideline Directed Medical Therapy (GDMT) Prescription in Heart Failure With Reduced Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOD00016877
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Patient Acceptance of Health Care
Keywords: heart failure with reduced ejection fraction; patient education
MeSH Terms: conditions — Heart Failure; Patient Acceptance of Health Care | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Intervention arm will receive initial face to face education during hospital admission and also an educational flier about GDMT. They will get 3 more sessions of education over phone at 1, 3 and 5 months after discharge, each session includes an overview of benefits and side effects of GDMT, inquiries about reasons of not using optimal doses of GDMT medications, and encouraging adherence to visits with providers.
  Interventions: Behavioral: Patient education
- Control (No Intervention): Control arm will receive initial face to face education during hospital admission and also an educational flier about GDMT.

INTERVENTIONS:
Behavioral: Patient education — 3 sessions of education over phone at 1, 3 and 5 months after discharge, each session includes an overview of benefits and side effects of GDMT, inquiries about reasons of not using optimal doses of GDMT medications, and encouraging adherence to visits with providers.
  Arms: Intervention

SUMMARY:
The goal of this randomized clinical trial is to test the effect of patient education on extent of use of guideline directed medical treatment (GDMT) of heart failure with reduced ejection fraction. The main question that our study aims to answer is if patient education can improve the adherence to GDMT in heart failure with reduced ejection fraction. Participants will receive educations about GDMT benefits in 1,3 and 5 months after discharge from hospital.

DETAILED DESCRIPTION:
This is a randomized clinical trial assessing the possible benefit of post-discharge education on the extent of guideline directed medical treatment for heart failure with reduced ejection fraction. Patients that are admitted to medical facilities of the Medstar health, Baltimore will be screened and if consented, they will all get an initial inhouse face to face education, and upon discharge, they will be randomized to the control group and intervention group. The latter will get more educations via phone-call sessions at 1, 3 and 5 months post discharge. The educational sessions will include educating the benefits of GDMT, reviewing the components of GDMT and their possible side effects, performing Medication reconciliation, Inquiries about reasons not getting the medications and encouraging adherence to clinic visits and requesting the treating providers for GDMT optimization. There will be no formal prescription or change of medication during the educational sessions. GDMT use will be assessed in all patients after 6 months according to GDMT score by the Heart Failure Collaboratory.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Heart Failure reduced Ejection Fraction (EF≤40%)
* Age >18 years
* Able to consent for enrollment.
* Hospitalized at one of the Medstar facilities (Inpatient)

Exclusion Criteria:

* Pregnancy
* Patient with stage D heart failure candidates for advanced therapies or on home inotropes or receiving hospice service
* Patients with advanced organ failure (End stage cancer, Advanced dementia, MELD (Model for End-Stage Liver Disease) score > 30, GFR (Glomerular filtration rate) <25) in whom GDMT is Futile
* Patients with Heart failure Collaboratory Score (HFCS) of 9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in GDMT score | 6 months
  Changes in GDMT score defined by the Heart Failure Collaboratory (Vericiguat and Ivabradine score will not be included in this study)

SECONDARY OUTCOMES:
Heart Failure hospitalization | 6 months
  Proportion of Heart failure hospitalization
cardiovascular death/Left Ventricular Assist Device implantation/Cardiac Transplant | 6 months
  Proportion of cardiovascular death/Left Ventricular Assist Device implantation/Cardiac Transplant
Number of GDMT classes of medications in use | 6 months
  Number of GDMT classes of medications in use

CONTACTS AND LOCATIONS:
Overall Officials: Anup Agarwal, MD, Principal Investigator — MedStar Health
Locations (4):
- United States (4):
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - Medstar Harbor Hospital, Baltimore, Maryland
  - Medstar Franklin Medical Center, Baltimore, Maryland
  - Medstar Good Samaritan Hospital, Baltimore, Maryland